CLINICAL TRIAL: NCT02662348
Title: T Cell Mediated Adaptive Therapy for Her2-positive Neoplasms of Digestive System
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yi Miao (Other)
Collaborators: Nanjing Abingen Biotech Co. Ltd (Other)
Responsible Party: Sponsor-Investigator, Yi Miao, Director of the Pancreas Research Centre; Director of Institute of Tumor Biology, Jiangsu Province Academy of Clinical Medicine, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-SR-116.F1
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Liver Cancer; Gallbladder Cancer; Bowel Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Gallbladder Neoplasms; Intestinal Neoplasms | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interleukin-2 Transfusion (Experimental): Patients receive low-dose Recombinant Human Interleukin-2 SC daily beginning 3 days before the first HER2Bi armed T cell infusions infusion.
  Interventions: Drug: Recombinant Human Interleukin-2
- T Cells Transfusion (Experimental): Patients receive HER2Bi-Armed T Cells IV weekly for 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: HER2Bi-Armed T Cells

INTERVENTIONS:
Drug: Recombinant Human Interleukin-2 — Given SC
  Other Names: Proleukin; Recombinant Human IL-2
  Arms: Interleukin-2 Transfusion
Drug: HER2Bi-Armed T Cells — Given IV
  Other Names: HER2Bi-Armed ATCs
  Arms: T Cells Transfusion

SUMMARY:
This phase I trial is to investigate the safety and the possible side effects of bi-specific antibody armed T-cell therapy when given together with low-dose IL-2 in treating patients with Her2-positive neoplasms of digestive system. Expanded autologues T cells that have been coated with bi-specific antibodies, such as anti-CD3 and anti-human epidermal growth factor receptor 2 (HER2), may stimulate the immune system in different ways and stop tumor cells from growing. Interleukin-2 may stimulate white blood cells to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Perform a phase I clinical trial to clearly define the toxicity profile of IV HER2Bi armed T cells in patients with neoplasms of digestive system.

SECONDARY OBJECTIVES:

I. Evaluate phenotype, cytokine profiles and tumor markers, cytotoxicity directed at laboratory Her2 positive cancer cell lines.

II. Evaluate the clinical symptoms and signs, clinical responses, imaging examination of pretherapy and post-treatment, cytokine profiles and tumor markers in serum before and after treatment, time to progression, and overall survival.

OUTLINE: This is a safety study of IV infused HER2Bi-armed activated T cells. Patients receive HER2Bi armed T cells IV weekly for 4 weeks. Patients also receive low-dose Interleukin subcutaneously (SC) daily beginning 3 days before the first HER2Bi armed T cells infusion. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with Her2-positive neoplasms of digestive system: IHC 3+
2. Clinical staging: Phase III or above
3. Ages: < 65
4. Expected survival time: > 1 year
5. Quality of Life: > 60
6. The functions of important organs( heart, liver, lung, kidney and etc.)are normal
7. The volunteers with informed consent

Exclusion criteria:

1. Patient with Her2-negative neoplasms of digestive system
2. Hepatic renal dysfunction
3. Cardiopulmonary insufficiency
4. Mental disorder
5. Allergic condition
6. With other malignant tumor
7. Lactating women
8. Patients with infection or received chemotherapy in the past two weeks
9. Patient with autoimmune disease using immunosuppressive drug
10. Patient with organ transplantation with long term use of immunosupresive drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by local and systemic toxicities | Up to 1 year

SECONDARY OUTCOMES:
Changes in cytokine profiles and tumor markers in serum before and after treatment | Baseline to up to 12 months
  Increases or decreases in the amount of cytokine produced from the pre-immunotherapy baseline at any time point after immunotherapy will be considered as continuous outcomes.
Changes in phenotyping induced by immunotherapy in peripheral blood mononuclear cells (PBMC) | Baseline to up to 12 months
  PBMC from the patients will be obtained before and after immunotherapy to determine if there are any phenotype changes induced by immunotherapy. Paired t-test will be used to compare the difference between baseline and after any time point of armed T cells treatment in T cell subpopulation (FACS), tumor marker (CBA/ELISA) and tumor killing ability of PBMC.
Clinical response rate (including clinical symptoms and signs, complete response, partial response, progressive disease, and stable disease, imaging examination of pretherapy and post-treatment) will be measured by follow-up investigation. | Up to 12 months
  Point and exact confidence interval estimates will be calculated for response rate.
Overall survival | Up to 12 months
  Will be estimated with the standard Kaplan-Meier method, from which summary statistics of interest (median, 6 month, 1-year rate, etc.) will be derived. Both point and 95% confidence interval estimates will be calculated.
Progression free survival | From the beginning of immunotherapy to progression or death, assessed up to 12 months
  Will be estimated with the standard Kaplan-Meier method, from which summary statistics of interest (median, 6 month, 1-year rate, etc.) will be derived. Both point and 95% confidence interval estimates will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Miao, PH.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Nov 2017 ( Anticipated)

REFERENCES:
- [Background] Molina MA, Codony-Servat J, Albanell J, Rojo F, Arribas J, Baselga J. Trastuzumab (herceptin), a humanized anti-Her2 receptor monoclonal antibody, inhibits basal and activated Her2 ectodomain cleavage in breast cancer cells. Cancer Res. 2001 Jun 15;61(12):4744-9. PMID 11406546
- [Background] Ross JS, Slodkowska EA, Symmans WF, Pusztai L, Ravdin PM, Hortobagyi GN. The HER-2 receptor and breast cancer: ten years of targeted anti-HER-2 therapy and personalized medicine. Oncologist. 2009 Apr;14(4):320-68. doi: 10.1634/theoncologist.2008-0230. Epub 2009 Apr 3. PMID 19346299
- [Background] Jorgensen JT. Targeted HER2 treatment in advanced gastric cancer. Oncology. 2010;78(1):26-33. doi: 10.1159/000288295. Epub 2010 Feb 25. PMID 20185938
- [Background] Camilleri-Broet S, Hardy-Bessard AC, Le Tourneau A, Paraiso D, Levrel O, Leduc B, Bain S, Orfeuvre H, Audouin J, Pujade-Lauraine E; GINECO group. HER-2 overexpression is an independent marker of poor prognosis of advanced primary ovarian carcinoma: a multicenter study of the GINECO group. Ann Oncol. 2004 Jan;15(1):104-12. doi: 10.1093/annonc/mdh021. PMID 14679128
- [Background] Janjigian YY, Werner D, Pauligk C, Steinmetz K, Kelsen DP, Jager E, Altmannsberger HM, Robinson E, Tafe LJ, Tang LH, Shah MA, Al-Batran SE. Prognosis of metastatic gastric and gastroesophageal junction cancer by HER2 status: a European and USA International collaborative analysis. Ann Oncol. 2012 Oct;23(10):2656-2662. doi: 10.1093/annonc/mds104. Epub 2012 Jun 11. PMID 22689179
- [Background] Takenaka M, Hanagiri T, Shinohara S, Kuwata T, Chikaishi Y, Oka S, Shigematsu Y, Nagata Y, Shimokawa H, Nakagawa M, Uramoto H, So T, Tanaka F. The prognostic significance of HER2 overexpression in non-small cell lung cancer. Anticancer Res. 2011 Dec;31(12):4631-6. PMID 22199341
- [Background] Mimura K, Kono K, Hanawa M, Kanzaki M, Nakao A, Ooi A, Fujii H. Trastuzumab-mediated antibody-dependent cellular cytotoxicity against esophageal squamous cell carcinoma. Clin Cancer Res. 2005 Jul 1;11(13):4898-904. doi: 10.1158/1078-0432.CCR-04-2476. PMID 16000588
- [Background] Pagni F, Zannella S, Ronchi S, Garanzini C, Leone BE. HER2 status of gastric carcinoma and corresponding lymph node metastasis. Pathol Oncol Res. 2013 Jan;19(1):103-9. doi: 10.1007/s12253-012-9564-2. Epub 2012 Aug 21. PMID 22907801
- [Background] Jorgensen JT, Hersom M. HER2 as a Prognostic Marker in Gastric Cancer - A Systematic Analysis of Data from the Literature. J Cancer. 2012;3:137-44. doi: 10.7150/jca.4090. Epub 2012 Mar 12. PMID 22481979
- [Background] Arnould L, Gelly M, Penault-Llorca F, Benoit L, Bonnetain F, Migeon C, Cabaret V, Fermeaux V, Bertheau P, Garnier J, Jeannin JF, Coudert B. Trastuzumab-based treatment of HER2-positive breast cancer: an antibody-dependent cellular cytotoxicity mechanism? Br J Cancer. 2006 Jan 30;94(2):259-67. doi: 10.1038/sj.bjc.6602930. PMID 16404427
- [Background] Hudis CA. Trastuzumab--mechanism of action and use in clinical practice. N Engl J Med. 2007 Jul 5;357(1):39-51. doi: 10.1056/NEJMra043186. No abstract available. PMID 17611206
- [Background] Krahn G, Leiter U, Kaskel P, Udart M, Utikal J, Bezold G, Peter RU. Coexpression patterns of EGFR, HER2, HER3 and HER4 in non-melanoma skin cancer. Eur J Cancer. 2001 Jan;37(2):251-9. doi: 10.1016/s0959-8049(00)00364-6. PMID 11166154
- [Background] Schuell B, Gruenberger T, Scheithauer W, Zielinski Ch, Wrba F. HER 2/neu protein expression in colorectal cancer. BMC Cancer. 2006 May 8;6:123. doi: 10.1186/1471-2407-6-123. PMID 16681853
- [Background] Kountourakis P, Pavlakis K, Psyrri A, Rontogianni D, Xiros N, Patsouris E, Pectasides D, Economopoulos T. Clinicopathologic significance of EGFR and Her-2/neu in colorectal adenocarcinomas. Cancer J. 2006 May-Jun;12(3):229-36. doi: 10.1097/00130404-200605000-00012. PMID 16803682
- [Background] Lum LG, Rathore R, Cummings F, Colvin GA, Radie-Keane K, Maizel A, Quesenberry PJ, Elfenbein GJ. Phase I/II study of treatment of stage IV breast cancer with OKT3 x trastuzumab-armed activated T cells. Clin Breast Cancer. 2003 Aug;4(3):212-7. doi: 10.3816/cbc.2003.n.028. No abstract available. PMID 14499016
- [Background] Davol PA, Smith JA, Kouttab N, Elfenbein GJ, Lum LG. Anti-CD3 x anti-HER2 bispecific antibody effectively redirects armed T cells to inhibit tumor development and growth in hormone-refractory prostate cancer-bearing severe combined immunodeficient beige mice. Clin Prostate Cancer. 2004 Sep;3(2):112-21. doi: 10.3816/cgc.2004.n.021. PMID 15479495
- [Background] Grabert RC, Cousens LP, Smith JA, Olson S, Gall J, Young WB, Davol PA, Lum LG. Human T cells armed with Her2/neu bispecific antibodies divide, are cytotoxic, and secrete cytokines with repeated stimulation. Clin Cancer Res. 2006 Jan 15;12(2):569-76. doi: 10.1158/1078-0432.CCR-05-2005. PMID 16428502
- [Background] Fu X, Tao L, Rivera A, Williamson S, Song XT, Ahmed N, Zhang X. A simple and sensitive method for measuring tumor-specific T cell cytotoxicity. PLoS One. 2010 Jul 29;5(7):e11867. doi: 10.1371/journal.pone.0011867. PMID 20686618
- [Background] Brown CE, Wright CL, Naranjo A, Vishwanath RP, Chang WC, Olivares S, Wagner JR, Bruins L, Raubitschek A, Cooper LJ, Jensen MC. Biophotonic cytotoxicity assay for high-throughput screening of cytolytic killing. J Immunol Methods. 2005 Feb;297(1-2):39-52. doi: 10.1016/j.jim.2004.11.021. Epub 2005 Jan 22. PMID 15777929
- [Background] Mann M, Sheng H, Shao J, Williams CS, Pisacane PI, Sliwkowski MX, DuBois RN. Targeting cyclooxygenase 2 and HER-2/neu pathways inhibits colorectal carcinoma growth. Gastroenterology. 2001 Jun;120(7):1713-9. doi: 10.1053/gast.2001.24844. PMID 11375952
- [Background] Zitron IM, Thakur A, Norkina O, Barger GR, Lum LG, Mittal S. Targeting and killing of glioblastoma with activated T cells armed with bispecific antibodies. BMC Cancer. 2013 Feb 22;13:83. doi: 10.1186/1471-2407-13-83. PMID 23433400
- [Background] Whenham N, D'Hondt V, Piccart MJ. HER2-positive breast cancer: from trastuzumab to innovatory anti-HER2 strategies. Clin Breast Cancer. 2008 Feb;8(1):38-49. doi: 10.3816/CBC.2008.n.002. PMID 18501058
- [Background] Ma J, Han H, Liu D, Li W, Feng H, Xue X, Wu X, Niu G, Zhang G, Zhao Y, Liu C, Tao H, Gao B. HER2 as a promising target for cytotoxicity T cells in human melanoma therapy. PLoS One. 2013 Aug 27;8(8):e73261. doi: 10.1371/journal.pone.0073261. eCollection 2013. PMID 24015299
- [Background] Zhang G, Liu R, Zhu X, Wang L, Ma J, Han H, Wang X, Zhang G, He W, Wang W, Liu C, Li S, Sun M, Gao B. Retargeting NK-92 for anti-melanoma activity by a TCR-like single-domain antibody. Immunol Cell Biol. 2013 Nov-Dec;91(10):615-24. doi: 10.1038/icb.2013.45. Epub 2013 Oct 8. PMID 24100387
- [Background] Han H, Ma J, Zhang K, Li W, Liu C, Zhang Y, Zhang G, Ma P, Wang L, Zhang G, Tao H, Gao B. Bispecific anti-CD3 x anti-HER2 antibody mediates T cell cytolytic activity to HER2-positive colorectal cancer in vitro and in vivo. Int J Oncol. 2014 Dec;45(6):2446-54. doi: 10.3892/ijo.2014.2663. Epub 2014 Sep 18. PMID 25242665
- [Background] Ma P, He Q, Li W, Li X, Han H, Jin M, Liu C, Tao H, Ma J, Gao B. Anti-CD3 x EGFR bispecific antibody redirects cytokine-induced killer cells to glioblastoma in vitro and in vivo. Oncol Rep. 2015 Nov;34(5):2567-75. doi: 10.3892/or.2015.4233. Epub 2015 Aug 28. PMID 26323605